CLINICAL TRIAL: NCT00571558
Title: Phase I Study of Photodynamic Therapy Using Pulsed Dye Laser and Oral Aminolevulinic Acid in Patients With Oral Leukoplakia
Brief Title: Photodynamic Therapy Using Aminolevulinic Acid in Treating Patients With Oral Leukoplakia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00842; NCI-2009-00842 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000579270; NU-NWU05-5-01 (Other: Robert H. Lurie Comprehensive Cancer Center); NWU05-5-01 (Other: DCP); P30CA060553 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2013-02

CONDITIONS: Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral | interventions — Aminolevulinic Acid; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

ARMS (1):
- Treatment (aminolevulinin acid and photodynamic therapy) (Experimental): Patients receive aminolevulinic acid PO 3-4 hours before undergoing photodynamic therapy using pulsed dye laser on day 1.
  Interventions: Drug: aminolevulinic acid hydrochloride; Drug: photodynamic therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: aminolevulinic acid hydrochloride — Given PO
  Other Names: 5-ALA HCl; ALA HCl; aminolevulinic acid HCl
Drug: photodynamic therapy — Undergo photodynamic therapy
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of photodynamic therapy using aminolevulinic acid in treating patients with oral leukoplakia. Photodynamic therapy uses a drug, such as aminolevulinic acid, that becomes active when it is exposed to a certain kind of light. When the drug is active, abnormal cells are killed. Photodynamic therapy using aminolevulinic acid may be effective against oral leukoplakia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity and feasibility of photodynamic therapy using pulsed laser therapy and oral aminolevulinic acid in treating patients with oral leukoplakia.

II. To define the dose-limiting toxicity and maximum tolerated dose of photodynamic therapy using pulsed laser therapy and oral aminolevulinic acid in these patients.

SECONDARY OBJECTIVES:

I. To assess the efficacy of photodynamic therapy using pulsed dye laser and oral aminolevulinic acid by examining clinical response at 1 and 3 months.

II. To determine quantitative histologic response at 3 months. III. To explore the association of response with specific molecular and biologic markers (i.e., DNA ploidy, proliferation using Ki-67, apoptosis using TUNEL, cyclin D1, and p53).

OUTLINE: This is a dose-escalation study of long pulsed dye laser light.

Patients receive aminolevulinic acid* orally (PO) 3-4 hours before undergoing photodynamic therapy using pulsed dye laser on day 1.

(Note: *Patients in cohort 1 and a latter cohort [to be determined during the course of the study] do not receive aminolevulinic acid before photodynamic therapy.)

Patients undergo biopsies of target lesions and clinically uninvolved mucosa 4-8 weeks before beginning therapy and then at 3 months for biomarker studies (DNA ploidy, p53, Ki-67, cyclin D1, and TUNEL assay). Blood is collected on days 1, 2, 14, 28, and 84 for toxicity assessment.

After completion of study treatment, patients are followed for up to 84 days.

ELIGIBILITY:
Criteria:

* Histologically confirmed oral leukoplakia with dysplasia OR oral leukoplakia with hyperplasia in a high-risk area (e.g., floor of mouth, tongue, or oropharynx)
* Multiple oral leukoplakia lesions are allowed however no more than 5 distinct lesions are biopsied and treated
* All lesions to be treated must be technically accessible by laser
* Patients with oral leukoplakia with hyperplasia in a non-high-risk location (e.g., buccal mucosa from ill-fitting dentures) are not allowed
* Must be willing to undergo baseline biopsies of leukoplakia lesion(s) and surrounding normal tissue 4-8 weeks before therapy and repeat biopsies at 3 months
* No evidence of ongoing radiation damage to the target site
* Karnofsky performance status (PS) 70-100% or Zubrod PS 0-1
* Life expectancy > 2 years
* Hemoglobin > 12 g/dL
* Platelet count > 100,000/mm^3
* ANC > 1,500/mm^3
* Creatinine =< 1.5 mg/dL
* SGPT and SGOT =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN (a higher level of bilirubin due to a familial metabolism will be considered on an individual basis)
* Willing to adhere to avoidance of sunlight and indoor light exposure for 24 hours after treatment
* Not pregnant or nursing
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to aminolevulinic acid
* No porphyria
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that, in the opinion of the investigators, would limit compliance or jeopardize the patient or integrity of the data
* Prior treatment for leukoplakia allowed
* No prior photodynamic therapy
* More than 3 months since prior participation in a clinical trial for leukoplakia
* More than 4 weeks since prior ablative therapy to the target lesion
* More than 4 weeks since prior and no concurrent psoralen or PUVA therapy
* No concurrent oral retinoids (e.g., isotretinoin)
* No concurrent use of tanning beds
* No other concurrent investigational agents
* Fertile patients must use effective contraception
* Patients with a previous diagnosis of stage I or II head and neck cancer are eligible provided definitive therapy, including radiation therapy, is completed and the patient has been rendered disease free for >= 2 years
* No chronic liver disease including those with normal liver function tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability with determination of optimal light dosing regimen, determination of dose limiting-toxicities, and maximum tolerated dose of photodynamic therapy using pulsed laser therapy and oral aminolevulinic acid | Up to 84 days

SECONDARY OUTCOMES:
Clinical response | 1 month
Clinical response | 3 months
Histologic response | 3 months
Mucosal risk marker modulation as measured by proliferation using Ki-67, apoptosis using TUNEL, cyclin D1, p53 expression, and DNA ploidy | Up to 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Wong Stuart, Principal Investigator — Robert H. Lurie Cancer Center
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin